CLINICAL TRIAL: NCT04888494
Title: Enhancing Cortical-hippocampal Functional Connectivity as a Novel Means for Relieving Chronic Low Back Pain
Brief Title: Hippocampal Stimulation in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Director Center for Translational Pain Research, Director Center of Excellence for Chronic Pain and Drug Abuse Research, Professor of Physiology, Anesthesia, PM&R Northwestern University, Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STU00211858; 5P50DA044121 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain; Back Pain; Pain
Keywords: transcranial magnetic stimulation; resting state MRI
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive the 2 modalities of stimulation (hippocampal and sham-TMS). Each stimulation round is composed by 5 daily sessions of stimulation, participants will not know which round is active and which is sham. The order of the stimulation modalities will be different across subjects. Subjects will be randomly assigned to one of two possible modality order according to the entrance in the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hippocampus-stimulation (Experimental): Active high-frequency rTMS (20 Hz pulse trains)
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham-stimulation (Experimental): Sham rTMS
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — For the brain stimulation the investigators will use Repetitive Transcranial Magnetic stimulation (rTMS). Different stimulation conditions (hippocampal or sham) will be delivered in each round of stimulation (5 days). Repetitive TMS will be applied at 100% resting motor threshold intensity, 20 Hz pulse trains separated by 28-s inter-train intervals (~20 minutes for the entire daily stimulation session). Stimulation parameters will be identical in both groups
  Arms: Hippocampus-stimulation
Device: Sham rTMS — Sham rTMS
  Arms: Sham-stimulation

SUMMARY:
In this study the investigators aim to examine the effects of Transcranial Magnetic Stimulation (TMS) on hippocampal network connectivity and pain levels in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months of back pain on a daily basis;
* male or female with no racial or ethnic restrictions;
* 18 to 75 years old;
* average back pain intensity > 4/10 at study entry;
* must be able to read, understand, and sign consent form;
* generally healthy.

Exclusion Criteria:

* back pain with fever, chills, rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures,
* history of tumor in the back;
* back surgery within the past 6 months;
* Chronic neurologic conditions, e.g., Parkinson's
* involvement in litigation regarding back pain;
* other severe medical diseases;
* pregnancy;
* positive urinary screen for any recreational drugs,
* opioids use;
* use of anticoagulants (low dose ASA allowed);
* history of gastric ulcer; renal insufficiency or congestive heart failure,
* contraindication to MRI,
* contraindication to TMS; including history of seizure/epilepsy*
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Diagnosis of major depression;
* Intra-axial implants (e.g. spinal cord stimulators or pumps)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Documents will be provided by Apkar Apkarian
Supporting Information: Study Protocol, ICF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened via a database maintained by one of the co-investigators. The first participant was enrolled on June 25, 2021, and the last participant was enrolled in February 2022.
Pre-assignment Details: Of the 44 participants screened, 16 met inclusion criteria and were randomized to treatment.
Groups:
- Hippocampus-stimulation First Then Sham-stimulation: Over five consecutive days, we use repetitive transcranial magnetic stimulation (rTMS) at the resting motor threshold intensity to stimulate a region of interest in the parietal cortex, which is determined based on its connectivity with the hippocampus. The rTMS consists of 1,600 pulses delivered in 2-second periods of 20 Hz pulse trains, with 28-second inter-train intervals. Each daily stimulation session lasts about 20 minutes.
  After a two-week washout period, we administer sham stimulation with identical parameters except that the coil is flipped over to the sham side, and a stimulating electrode is attached to the skin near the parietal rTMS target location. This electrode delivers a small current to mimic the physical sensation of real stimulation, making it difficult for participants to discriminate between the two types of stimulation.
- Sham-stimulation First Then Hippocampus-stimulation: For five consecutive days, we administer sham stimulation by flipping the coil over to the sham side and attaching a stimulating electrode to the skin near the parietal rTMS target location. The electrode delivers a small current to mimic the physical sensation of real stimulation, making it difficult for participants to distinguish between the two types of stimulation. Each daily stimulation session lasts around 20 minutes.
  After a two-week washout period, we use repetitive transcranial magnetic stimulation (rTMS) at the resting motor threshold intensity to stimulate a region of interest in the parietal cortex, which will be determined based on its connectivity with the hippocampus. The rTMS consists of 1,600 pulses delivered in 2-second periods of 20 Hz pulse trains, with 28-second inter-train intervals.
Period: Overall Study
Arm/Group | Hippocampus-stimulation First Then Sham-stimulation | Sham-stimulation First Then Hippocampus-stimulation
Started | 8 | 8
First Intervention (5 Days) | 5 | 5
Washout (14 Days) | 5 | 5
Second Intervention (5 Days) | 5 | 5
Completed | 5 | 5
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — We dropped the participant due to safety concerns for the staff. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hippocampus-stimulation First, Then Sham-stimulation: Over five consecutive days, we use repetitive transcranial magnetic stimulation (rTMS) at the resting motor threshold intensity to stimulate a region of interest in the parietal cortex, which is determined based on its connectivity with the hippocampus. The rTMS consists of 1,600 pulses delivered in 2-second periods of 20 Hz pulse trains, with 28-second inter-train intervals. Each daily stimulation session lasts about 20 minutes.
  After a two-week washout period, we administer sham stimulation with identical parameters except that the coil is flipped over to the sham side, and a stimulating electrode is attached to the skin near the parietal rTMS target location. This electrode delivers a small current to mimic the physical sensation of real stimulation, making it difficult for participants to discriminate between the two types of stimulation.
- Sham-stimulation Then Hippocampus Stimulation: For five consecutive days, we administer sham stimulation by flipping the coil over to the sham side and attaching a stimulating electrode to the skin near the parietal rTMS target location. The electrode delivers a small current to mimic the physical sensation of real stimulation, making it difficult for participants to distinguish between the two types of stimulation. Each daily stimulation session lasts around 20 minutes.
  After a two-week washout period, we use repetitive transcranial magnetic stimulation (rTMS) at the resting motor threshold intensity to stimulate a region of interest in the parietal cortex, which will be determined based on its connectivity with the hippocampus. The rTMS consists of 1,600 pulses delivered in 2-second periods of 20 Hz pulse trains, with 28-second inter-train intervals.
- Total: Total of all reporting groups
Arm/Group | Hippocampus-stimulation First, Then Sham-stimulation | Sham-stimulation Then Hippocampus Stimulation | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (18) | 52 (15) | 55 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Baseline Pain [Mean (Standard Deviation); unit: units on a scale] — The severity of baseline pain is measured with the Numeric Rating Scale (NRS) scores. The NRS is a pain screening tool that assesses pain severity during assessment using a 0-10 scale, where zero means "no pain" and ten means "the worst pain imaginable."
  units on a scale | 4.6 (1.9) | 4.6 (1.8) | 4.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Pain Scales
Description: The endpoint will be the severity of pain measured by changes in the Numeric Rating Scale (NRS) scores before and after each stimulation round. The NRS is a pain screening tool that assesses pain severity during assessment using a 0-10 scale, where zero means "no pain" and ten means "the worst pain imaginable." Higher values indicate a worse outcome.
Time Frame: Pain is assessed at baseline, end of first intervention and end of the second intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hippocampus-stimulation: Over five consecutive days, we use repetitive transcranial magnetic stimulation (rTMS) at the resting motor threshold intensity to stimulate a region of interest in the parietal cortex, which is determined based on its connectivity with the hippocampus. The rTMS consists of 1,600 pulses delivered in 2-second periods of 20 Hz pulse trains, with 28-second inter-train intervals. Each daily stimulation session lasts about 20 minutes.
- Sham-stimulation: For five consecutive days, we administer sham stimulation by flipping the coil over to the sham side and attaching a stimulating electrode to the skin near the parietal rTMS target location. The electrode delivers a small current to mimic the physical sensation of real stimulation, making it difficult for participants to distinguish between the two types of stimulation. Each daily stimulation session lasts around 20 minutes.
Arm/Group | Hippocampus-stimulation | Sham-stimulation
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 4.6 (1.9) | 4.6 (1.9)
  After Intervention | 4 (2.2) | 4.4 (1.8)

2. Secondary Outcome: Changes in Hippocampal Connectivity
Description: Changes in hippocampal network connectivity will be evaluated by using resting state functional magnetic resonance (fMRI) before and after hippocampal stimulation. Hippocampal connectivity measurements - regions involved in the network and the parietal target - will be compared before stimulation (baseline) to after stimulation (after active hippocampal stimulation).
Time Frame: approximately 6 weeks - Baseline and after the end of hippocampal stimulation
Population: The data was not collected due to the COVID-19 pandemic.
Arm/Group | Hippocampus-stimulation First, Then Sham-stimulation | Sham-stimulation Then Hippocampus Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every visit (protocol) through study completion, an average of seven weeks
Groups:
- Hippocampus-stimulation: Different stimulation conditions (hippocampal or sham) will be delivered in each round of stimulation (5 days). Repetitive TMS will be applied at 100% resting motor threshold intensity to a region of interest located in the parietal cortex, which will be determined based on its connectivity with the hippocampus. This stimulation consists of a series of 1,600 pulses administered as 2-second periods of 20 Hz pulse trains separated by 28-s inter-train intervals (~20 minutes for the entire daily stimulation session).
- Sham-stimulation: Parameters will be identical to the hippocampus-stimulation, except that the coil will be flipped over to the sham side, and a stimulating electrode will be attached to the skin near the parietal rTMS target location. This electrode will be used to deliver a small current mimicking real stimulation sensation; therefore, participants cannot reliably discriminate physical sensations for real versus sham rTMS.
Arm/Group | Hippocampus-stimulation | Sham-stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04888494/Prot_SAP_000.pdf